CLINICAL TRIAL: NCT05051657
Title: A Study To Evaluate The Acceptability Of the Express Plus Range, Foods For Special Medical Purposes (FSMP), In Children And Adults With Inborn Errors of Metabolism (IEM)
Brief Title: Evaluation of the Express Plus Range
Acronym: express plus
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vitaflo International, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCT-EXPP-2019-05-21; 281995 (Other: IRAS); 20/YH/0248 (Other: Sheffield Research Ethics Committee)
Record Dates: First submitted 2021-09-10; First posted 2021-09-21 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Phenylketonurias; PKU; Homocystinuria; Maple Syrup Urine Disease; Hereditary Tyrosinemia; Glutaric Acidemia I
MeSH Terms: conditions — Phenylketonurias; Homocystinuria; Maple Syrup Urine Disease; Tyrosinemias; Glutaric Acidemia I

STUDY DESIGN:
Intervention Model Description: single group - all patients to receive relevant express plus product
Masking Description: No masking, product will be given open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- express pus range (PKU, MSUD, HCU, TYR and GA) (Experimental): express plus to be transitioned onto over a maximum of 6 weeks and then incorporated into each participants usual diet for 28 days. Amount taken and frequency to be determined by dietitian.
  Interventions: Dietary Supplement: PKU express plus

INTERVENTIONS:
Dietary Supplement: PKU express plus — PKU express plus is a powdered protein substitute for the dietary management of PKU. It is formulated in a variety of flavours to provide a convenient, low volume, lower calorie, pre-measured protein substitute, containing a full micronutrient profile.

SUMMARY:
A prospective, open label, acceptability study to evaluate PKU, MSUD, HCU, TYR and GA express plus in the dietary management of 40 patients with IEM. The following parameters will be assessed: adherence to prescribed dietary intakes, palatability, usability, gastrointestinal tolerance, clinically relevant routine biochemical parameters, timeframe to transition and contribution of the express plus range to overall protein substitute intake over a 28 day period.

DETAILED DESCRIPTION:
This is a prospective acceptability study of the express plus range in 40 participants aged at least three years of age for the dietary management of IEM (PKU, MSUD, HCU, TYR and GA ).

The study will involve a Transition Period where patients will build-up to at least one sachet of express plus per day. During the Transition Period, daily intake of express plus and the patient's other PS will be recorded, including the time taken to consume.

The Transition Period will last a maximum of 6 weeks, after which the patient will enter a 28-day Evaluation Period. During the Evaluation Period, patients will continue to record intakes, as well as GI tolerance and a final evaluation of the product's palatability and usability. Some patients, likely adults, will not require a transition from their original protein substitute to at least one sachet of express plus. These patients can enter the Evaluation Period directly.

The end of the 4-week Evaluation Period is defined as the participant's End of Study. Following this, participants will be followed up as per standard of care. Some of this standard of care data may be relayed to the sponsor for a maximum of 26 weeks. This will last for a maximum of 26 weeks and will involve the collection of routine phe and tyrosine levels, as well as amount of PS prescribed and taken. Information will also be collected from patients regarding the reasons for the success or indeed failure of transition to PKU express plus. This data will come from routine clinical contact and will be recorded by the HCP, rather than by the patient.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PKU or associated disorder for example, Tetrahydrobiopterin (BH4) deficiency, requiring a low protein diet and Phe-free L-amino acid supplements (protein substitute).
* Established on PKU express or an equivalent protein substitute
* In the opinion of the study investigator, the participant is able to take the study product and meets at least one of the following criteria:

  1. taking an age inappropriate protein substitute
  2. struggling with adherence to current protein substitute
  3. delayed in transitioning
* Aged 3 years and above
* Willingly given, written, informed consent from patient or parent/guardian.
* Willingly given, written assent (if appropriate).

Exclusion Criteria:

* Diagnosis of persistent hyperphenylalaninaemia, or mild PKU not requiring dietary intervention with a low protein diet and protein substitute.
* Patients who are tube-fed.
* Individuals, who in the opinion of the investigator, are unable to comply with the requirements of the protocol.
* Any co-morbidity/condition which in the opinion of the Investigator, would preclude participation in the study.
* Patients who are currently participating in, plan to participate in, or have participated in an interventional investigational drug, food or medical device trial within 30 days prior to screening.
* Use of additional macro/micronutrient supplements during the study period, unless clinically indicated and prescribed by the investigator (must be recorded in patient case record file).
* Women who are pregnant / breastfeeding at the start of the study or planning to become pregnant during the study period. (N.B.: Women who become pregnant unexpectedly during this study may, in consultation with their doctor, continue on the study's dietary product if they wish but will not have any investigations that would not normally be carried out during pregnancy.)
* Those with allergies to fish, milk or soya.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Questionnaire of self-reported adherence to the prescribed amount of study product | Days 1-28
  Participants will record the amount of PKU express taken each day compared to the amount recommended by their dietitian
Transition time | Transition period Weeks 1-6 (maximum)
  Time taken for participants to transition from their current diet to the inclusion of one sachet of PKU express plus per day
Change in gastrointestinal tolerance from week 1 to week 4 | Days 1-7 and days 21-28
  Participants will self-report any gastrointestinal symptoms experience over the course of the study in daily study diaries
Product acceptability rated on a Likert scale by the patient after 28-day intake | Visit 2 (end of 28 day evaluation period)
  Participants will answer questions relating to PKU express plus' palatability and ease of use following the end of study
Change in general neophobia | Visit 1 (Day 1) and Visit 2 (end of 28 day evaluation period)
  Participants to complete general neophobia questionnaire at baseline and end of study to compare results
Change in food neophobia | Visit 1 (Day 1) and Visit 2 (end of 28 day evaluation period)
  Participants to complete food neophobia questionnaire at baseline and end of study to compare results
Nutritional suitability: change Phenylalanine levels | Visit 1 until visit 2 (day 28)
  PKU express plus' nutritional suitability will be assessed by evaluating Phenylalanine levels recorded as part of routine care
Nutritional suitability: change Tyrosine levels | Visit 1 until visit 2 (day 28)
  PKU express plus' nutritional suitability will be assessed by evaluating Tyrosine levels recorded as part of routine care

CONTACTS AND LOCATIONS:
Overall Officials: Anita MacDonald, Study Director — Birmingham Women's and Children's Hospital
Locations (6):
- United Kingdom (6):
  - Royal Belfast Hospital for Sick Children, Belfast
  - Birmingham Women's and Children's Hospital, Birmingham
  - Bristol Royal Hospital for Children, Bristol
  - Greater Glasgow and Clyde NHS Foundation Trust, Glasgow
  - Great Ormond Street Hospital for Children, London
  - Nottingham Children's Hospital, Nottingham

IPD SHARING:
Plan to Share IPD: No
No plans to share IPD